CLINICAL TRIAL: NCT00774085
Title: Electronic Schizophrenia Treatment Adherence Registry
Brief Title: An Observational Study to Assess Treatment & Outcomes Data in Patients Receiving Long-Acting Injectable Risperidone
Acronym: e-STAR
Status: Completed | Type: Observational
Sponsor: Janssen Cilag N.V./S.A. (Industry)
Responsible Party: SR MEDICAL ADVISOR, Jan-Cil Benelux
Other Study IDs: CR003886; RISSCH4002 (Other: Janssen Cilag N.V./S.A., Belgium); 2004-002448-93 (EudraCT Number)
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Risperidone; Risperdal Consta; Propective; Retrospective; Mental disorders; Observational
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with Schizophrenia: Patients with Schizophrenia are treated with long-acting injectable risperidone (Risperdal Consta) in daily practice according to local label by the physicians
  Interventions: Other: No intervention was given

INTERVENTIONS:
Other: No intervention was given — Participants included patients treated with long-acting injectable risperidone (Risperdal Consta) in daily practice according to local label by the physicians

SUMMARY:
The purpose of this study is to assess treatment and outcomes data in patients receiving treatment with long-acting injectable risperidone.

DETAILED DESCRIPTION:
This is an observational (study in which patients/participants are observed) and multicentre (at multiple sites) study. This is one-country arm of a multinational study. This study consists of 2 years of retrospective (a study in which the patients are identified and then documented backward in time and 2 years of prospective (a study in which the patients are identified and then followed forward in time for the outcome of the study) study periods during which medication utilization review will be done, determining medication usage patterns and outcomes associated with the use of risperidone long acting, in clinical practice. Usage of risperidone according to label was recommended during the study. The planned recruitment period will be 6 months. Retrospective observation will be 2 years for hospitalization history and at least 1 year for medication usage. Total duration of prospective observation for each patient with a complete follow-up will be 24 months. Data collection during the follow up period will be scheduled every 3 months ± 2 weeks. In addition, this study is proposed in Belgium to satisfy the demand from Belgian Reimbursement Authorities to collect clinical data on the impact of risperidone long acting on treatment compliance, number of hospitalizations and potential prevention of relapses. Also, this data will provide documentation on switch from oral to parenteral treatment. Data will be pooled from different physicians and/or countries. The objectives of this study are: collect clinical outcome data at the request of the Belgian Reimbursement Authorities; prospectively assess medication usage patterns to document clinical efficacy and long-term treatment outcomes of risperidone long acting, in a naturalistic setting; collect retrospective data, to compare with risperidone long acting; document reasons for initiating risperidone; collect data on switch of treatment to risperidone long acting.

ELIGIBILITY:
Inclusion Criteria:

* Patient who started long-acting injectable risperidone treatment after agreement between doctor and patient
* Ambulatory patient or not chronically full-time hospitalized patient. Full-time hospitalization at the moment of inclusion for maximal 6 months
* The treatment and treated indication according to local label
* Patient had given informed consent in agreement with local legislation

Exclusion Criteria:

* Patient participating in another medication related study, chronically full-time hospitalized patient, who according to the treating physician had no perspective of being discharged within the planned observation period
* Patient suffering from treatment resistant schizophrenia
* Pregnant or breastfeeding females or females with planned pregnancy within two years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with schizophrenia
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2004-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in total length of hospitalization from retrospective to prospective period | 48 months
  Start date, end date of full-time or partial hospitalization will be recorded both in retrospective and prospective study period.

SECONDARY OUTCOMES:
Change from baseline to 24 months in Clinical Global Impression (CGI) Scale scores | Baseline, (just before the first injection of long-acting injectable risperidone) to 24 months
  Patients are rated for overall severity of schizophrenia disorder using the CGI scale (7 point scale) in which 1 = Not Ill and 7 = Extremely Severe.
Change from baseline to 24 months in Global Assessment of Functioning (GAF) scores | Baseline to 24 months
  This GAF scale rates the functioning of the patient on a scale of 1 - 100 where "1 - 10" is "Persistant danger of severely hurting self or others (eg, recurrent violence) OR persistant inability to maintain personal hygiene OR serious suicidal act with clear expectations of death" and "91- 100" is "Superior functioning in a wide range of activities, life's problems never seem to get out of hand, is sought out by others because of his of her positive qualities. No symptoms"
Change from baseline to 24 months in clinical deterioration | Baseline, in 3-monthly intervals (± 2 weeks) for 24 months and Last visit
  Clinical deterioration is assessed by evaluating presence or absence of deliberate self injury, suicidal or homicidal ideation, violent behaviour, and increased need in levels of care and increase in CGI by 2 points or more. The maintenance of treatment effect is documented by the time to significant deterioration of the psychotic condition. If signs of significant deterioration occurred more than once within each 3 monthly interval, this is recorded.
Change from baseline to 24 months in assessment of remission | Baseline to 24 months
  Clinical status will be assessed by presence or absence of the following core symptoms: delusions, conceptual disorganization, hallucinatory behavior, mannerisms and posturing, unusual thought content, blunted affect, passive/apathetic social withdrawal, lack of spontaneity and flow of conversation. Score will be given for each symptom as follows: Score 1: Absent, Minimal, Mild; Score 2: Moderate, Moderately severe, Severe, Extreme. Symptomatic remission is defined as a clinical status where for each and every of the symptoms prespecified, a score of 1 can be given for duration of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag N.V./S.A., Belgium Clinical Trial, Study Director — Janssen Cilag N.V./S.A.